CLINICAL TRIAL: NCT04779086
Title: Investigation of E-health Literacy Levels of Physiotherapy and Rehabilitation Department Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Rabia Tugba Kilic, Assistant Professor, Ankara Yildirim Beyazıt University
Other Study IDs: 2020-282
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Health Behavior; Health Attitude; Health Knowledge
Keywords: e-health literacy, physiotherapy and rehabilitation
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1. group: Scale score results of first year physiotherapy and rehabilitation department students
- 2. group: Scale score results of 2nd year physiotherapy and rehabilitation department students
- 3. group: Scale score results of 3rd year physiotherapy and rehabilitation department students
- 4. group: Scale score results of 4th year physiotherapy and rehabilitation department students

SUMMARY:
This study will be carried out in order to determine the e-health literacy levels of the students of the Department of Physiotherapy and Rehabilitation and to reveal whether the level of their education has an effect on e-health literacy.

It is aimed to contribute to the literature with the objective, evidence-based results to be obtained from the study and to contribute to undergraduate education as a result of the differences between class levels.

DETAILED DESCRIPTION:
Health literacy is generally affected by many factors, from demographic, cultural and psychosocial factors, general literacy level, individual characteristics, experiences related to the disease, and factors related to the healthcare system. It is stated that the evidence supporting the negative effects on the health of individuals is increasing due to the lack of health literacy.

These effects; Low use of preventive healthcare services are shown as delay in seeking health care in the symptomatic period, inability to understand the medical condition of the individual, inability to adhere to medical advice / instructions, insufficient self-care, increase in health care costs and increase in mortality.

In terms of health, health literacy is a stronger determinant than income, employment status, education level, race or ethnic group . The strong place of the concept of health literacy among the main determinants of health appears to be an important factor in the struggle for inequality in health. It is stated that adoption of lifelong learning policies to increase health literacy has important effects .

Since health literacy is directly related to general literacy, studies to be carried out in the field of education can contribute to health literacy and to the improvement of health, thereby reducing health inequalities. It has been determined that the e-health literacy levels of the students studying at Kırıkkale University Faculty of Health Sciences in 2016-2017 differ according to the departments, they are at medium and high levels (average 29.48).

Studies have been suggested to improve the e-health literacy levels of Faculty of Health Sciences students. These recommendations are in line with this study is to determine the students of Physiotherapy and Rehabilitation Department e-health literacy levels in Turkey and will be conducted to determine whether there is effective on the e-health literacy attended class. In case of a difference, secondary goal is to improve the level of health literacy by contributing to undergraduate education.

ELIGIBILITY:
Inclusion Criteria:

* 1st, 2nd, 3rd and 4th year students studying in the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences in 2020-2021
* Volunteer to participate in the study

Exclusion Criteria:

* Those who do not study at the Faculty of Health Sciences, Physiotherapy and Rehabilitation Department of universities
* Not volunteering to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1st, 2nd, 3rd and 4th year students studying in the Department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences in 2020-2021 and; The data will be obtained from the students who agree to participate in the study by using a questionnaire method.
Sampling Method: Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
E-health Literacy Levels | 5 months
  E-health Literacy E-health Literacy scale score,The scale score is a minimum of 8 and a maximum of 40 points. The higher the score, the higher the health literacy level.

CONTACTS AND LOCATIONS:
Overall Officials: Rabia Tugba Kilic, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University,Faculty of Health Sciences, Physiotherapy and Rehabilitation Department, Ankara, Turkey (Türkiye)

REFERENCES:
- [Result] Sorensen K, Van den Broucke S, Fullam J, Doyle G, Pelikan J, Slonska Z, Brand H; (HLS-EU) Consortium Health Literacy Project European. Health literacy and public health: a systematic review and integration of definitions and models. BMC Public Health. 2012 Jan 25;12:80. doi: 10.1186/1471-2458-12-80. PMID 22276600
- [Result] Whitehead M, Dahlgren G. What can be done about inequalities in health? Lancet. 1991 Oct 26;338(8774):1059-63. doi: 10.1016/0140-6736(91)91911-d. No abstract available. PMID 1681366
- [Result] Kickbusch IS. Health literacy: addressing the health and education divide. Health Promot Int. 2001 Sep;16(3):289-97. doi: 10.1093/heapro/16.3.289. PMID 11509466
- [Result] Bilir LK. Patent laws, product life-cycle lengths, and multinational activity. American Economic Review. 2014;104(7):1979-2013.
- [Result] Yılmaz A, Saygılı M, Kaya M. Sağlık Bilimleri Fakültesi Öğrencilerinin E-Sağlık Okuryazarlığı Düzeylerinin Belirlenmesi. Mehmet Akif Ersoy Üniversitesi Sosyal Bilimler Enstitüsü Dergisi. 2020 (May) : 31.
- [Result] Norman CD, Skinner HA. eHEALS: The eHealth Literacy Scale. J Med Internet Res. 2006 Nov 14;8(4):e27. doi: 10.2196/jmir.8.4.e27. PMID 17213046
- [Result] Coşkun S, Bebiş H. Psychometric evaluation of a Turkısh version of the e-health literacy scale (e-heals) in adolescent. Gülhane Tip Dergisi. 2015;57(4):378.